CLINICAL TRIAL: NCT06178237
Title: RADA16 for Reducing Drain Output Trajectory Following Neck Dissection
Acronym: ROUND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. James's Hospital, Ireland (Other)
Collaborators: Royal College of Surgeons, Ireland (Other)
Responsible Party: Principal Investigator, Gerard Sexton, Specialist Registrar in Otolaryngology, St. James's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 000117
Record Dates: First submitted 2023-10-31; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancer
Keywords: seroma
MeSH Terms: conditions — Head and Neck Neoplasms; Seroma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Standard of care post-neck dissection
- Standard of care plus Purabond (Experimental): Standard of care post-neck dissection plus Purabond
  Interventions: Device: Purabond

INTERVENTIONS:
Device: Purabond — Application of Purabond to surgical field
  Other Names: RADA16
  Arms: Standard of care plus Purabond

SUMMARY:
This will be a prospective single-blind randomised controlled trial to evaluate if the use of a medical device named Purabond, a haemostatic agent already CE marked for use in Ireland, can reduce the occurrence of seroma, a complication related to but distinct from haematoma, following neck dissection surgery. Patients undergoing neck dissection surgery will be randomised either to standard post-operative care following neck dissection or to standard post-operative care and Purabond. Drains are placed routinely following surgery of this type and their removal is dictated by the volume of fluid produced per day - it is hypothesised that Purabond will reduce the volume of fluid produced and thereby facilitate earlier drain removal.

DETAILED DESCRIPTION:
Purabond is a new medical device taking the form of a gel containing an active ingredient called RADA-16. It is designed to stop bleeding from wounds by forming into a stable barrier (matrix) when coming into contact with ionic fluids like blood. Purabond is already currently use for procedures by Cardiology, General Surgery, Vascular, Gynaecology, and ENT. Specific uses in ENT surgery so far have been for sinus surgery. Purabond is CE marked and indicated for situations where haemostasis by standard means is insufficient or impractical.

The investigators hypothesise that Purabond will reduce the duration for which neck drains must be left in place after neck dissection, which is an operation to remove lymph nodes from the neck. Following neck dissection, fluid can leak into the healing tissues in the neck from very small damaged blood vessels - when an excess of this fluid builds up underneath the skin this is called a seroma. This occurs in 1.3-7% of patients and represents a potential area for infection as well as a noticeable lump. Readmission is sometimes required in the event of an infected seroma though there is no published evidence on how common this is. Drains are placed during neck dissection surgery to remove this fluid and to also reduce the overall seroma rate. Drains are left in until the volume of fluid being produced decreases. The duration for which drains are left in place is also affected by the development of other, rarer complications - specifically chyle leak, anastomotic leak, and pharyngocutaneous fistula. In the setting of any of the above, drains are often left in for longer to ensure any fluid that accumulates is removed and that dead space in the neck is kept to a minimum.

This study aims to assess if Purabond can speed up the process of removing drains. The fluid that makes up a seroma leaks out from damaged blood vessels in the same way a haematoma (collection of blood in the neck) does but the vessels of interest in a seroma are smaller and more numerous - manual ligation of these is not feasible. As Purabond forms a matrix in response to ionic fluids (including seroma) it is expected to reduce the rate of seroma by sealing such vessels. The benefits of this would be reduced duration of stay in hospital for patients with otherwise uncomplicated neck dissections but also reducing infection risk to patients with more complex needs who could otherwise have their drains removed earlier. It would also be expected to reduce the subsequent need for readmission and aspiration of seroma. These findings would then be more broadly applicable to less extensive neck surgeries where there is a risk of seroma but drains are not placed frequently (parotidectomy, thyroidectomy, etc).

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck cancer (including thyroid, cutaneous, & mucosal primaries) for which a neck dissection is indicated as part of treatment.
* Over 18 years of age.
* Able to give informed consent.

Exclusion Criteria:

* Patients unable to satisfy all the above listed inclusion criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Total volume of fluid drained | 3 months
  Total output from intraoperatively placed drain plus any additional drainage performed percutaneously
Duration of drain placement | Until drain removal, usually within 2 weeks
  Duration of drain placement

SECONDARY OUTCOMES:
Haematoma | Usually within 1 week
  Haematoma
Number of percutaneous aspirations required | 3 months
  Number of percutaneous aspirations required
Duration of inpatient stay | 3 months
  Duration of inpatient stay
Number of patients with neck dissection complications relevant to drains management | 3 months
  Complications affecting drain management - chyle leak, pharyngocutaenous fistula, anastomotic leak

IPD SHARING:
Plan to Share IPD: Undecided